CLINICAL TRIAL: NCT00521534
Title: Impact of Resynchronization Therapy on Sleep Disordered Breathing in Advanced Congestive Heart Failure
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Collaborators: Boston Scientific Corporation (Industry); University of Pittsburgh (Other)
Responsible Party: Alaa Shalaby, MD, VA Pittsburgh Healthcare System
Other Study IDs: 02345
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Sleep Related Breathing Disorder; Congestive Heart Failure
Keywords: Sleep related Breathing Disorder; Congestive Heart Failure; Atrial Overdrive Pacing; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: CRT programmed to VDD pacing mode
- B: CRT programmed to DDD with overdrive pacing based on first night average sinus rate.
  Interventions: Device: CRT with atrial overdrive pacing

INTERVENTIONS:
Device: CRT with atrial overdrive pacing — Both groups receive CRT, one group receives atrial overdrive pacing
  Groups: B

SUMMARY:
Background and Introduction:

SDB is increasingly recognized as a co-morbidity with significant impact on overall health. The disorder has been implicated in the development of hypertension, atherosclerotic cardiovascular disease as well as arrhythmia, stroke and the progression of congestive heart failure. The disorder is prevalent among males, estimated to affect upto 24% of the general population. Its prevalence increases with age, and it is particularly prevalent among patients with congestive heart failure with the prevalence rising to 51% in that group. Interestingly, recent evidence points to a potential impact for treating sleep disordered breathing, on heart failure patients. At the same time, recent reports of a beneficial impact of atrial overdrive pacing on SDB, have stirred interest in a potentially effective and well tolerated non-pharmacologic means of therapy for this disorder. Particularly at a time when cardiac resynchronization therapy utilizing biventricular pacing has demonstrated significant impact on heart failure, the interplay between CHF and SDB pacemaker based therapy begs further exploration. The interdependence of potential positive impact on each entity needs to be elucidated for further research and refinement of therapeutic tools. Furthermore, this study aims to explore potential neurohormonal influence on and affection by each of these disorders.

Specific Aims and Hypotheses:

Specific Aim #1: To assess the effect of cardiac resynchronization therapy (CRT) with or without atrial pacing on SDB in patients with advanced CHF at 8 and 16 weeks after implementation of therapy.

Hypothesis #1: Resynchronization therapy improves SDB, the effect may anticipate or lag improvement in heart failure. Atrial pacing has a beneficial effect in addition to CRT.

Specific Aim #2: To explore the effect of CRT on cardiac neuro-hormonal activity in relation to its effects on CHF and SDB.

Hypothesis #2: CRT neuro-hormonal modulation is a common path in its effects on SDB and CHF.

Specific Aim #3: To assess prevalence of sleep disordered breathing (SDB) in patients with advanced congestive heart failure (CHF).

Hypothesis #3: SDB is prevalent yet under recognized in this patient population.

Research Design:

This is an observational study with a built in double blinded prospective randomized interventional substudy of a potential confounder i.e. atrial pacing. All patients will receive CRT with defibrillator for clinical indications (CRT-D). Investigators other than the EP physicians as well as patients will be blinded to the pacing mode. After screening and a run in period of back up pacing a baseline polysomnogram (PSG) will be performed. Patients will be randomized between atrial overdrive or atrial tracking pacing modes for six months, all patients receiving CRT. Sleep studies will be performed at baseline and at three month intervals. Subjects: Patients referred for implantation of CRT -D will be recruited for this trial. Patients are included only if they are indicated for such a device on clinical grounds. Outcome Measures: 1.Sleep quality related Parameters:The following will be collected at times of each PSG: MAP-PSQI, PSG parameters of sleep quality and architecture, apnea hypopnea index, and oxygen saturation as well as biochemical markers of sleep efficiency. 2.Heart Failure Parameters: The following will be obtained at times of each PSG: Minnesota Living with Heart Failure Questionnaire, Clinical and echocardiographic measures of heart failure progression and biochemical markers of heart failure severity.

Power Analysis: An improvement in SDB in both initial randomization arms is assumed, however we further assume the atrial overdrive arm will offer improvement over the atrial tracking arm of equal magnitude. An arbitrary estimate would be twenty percent improvement in atrial overdrive arm. The corresponding estimate is 40% improvement due to CRT. To achieve 0.80 power thirty four data sets need to be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18years
* Indication for CRT device implant:

  * Congestive heart failure (NYHA Class III or IV)
  * Ejection fraction less than 36%
  * Evidence of intraventricular dyssynchrony (QRS duration >120ms or positive tissue doppler echocardiogram).
  * Have a life expectancy of at least 6 months
  * Are on optimal pharmaceutical therapy (OPT)
* Ability and willingness to sign informed consent

Exclusion Criteria:

* Unstable angina, Canadian Cardiac Society Class III or greater.
* Patients with unstable heart failure defined as need for intravenous inotropes or inability to achieve stable medical regimen for 48 hours.
* Deterioration in CHF at any time during the study requiring hospital admission and any of the following:

  * A significant change in pharmaceutical regimen (see below: Pharmacologic Therapy)
  * A change in pacing mode parameters (with the exception of if the mode is inadvertently programmed incorrectly at implant)
  * A need for inotrope support
  * A downward change in functional class by one grade at discharge
* Women of childbearing age who are pregnant or who refuse pregnancy test and reliable contraception means for the duration of the study.
* Not having a successful percutaneous CRT device implant.
* Chronic atrial fibrillation.
* Patients currently known to have sleep apnea for which they are being treated with CPAP. (Patients prescribed to CPAP who have not been compliant for one month or greater are eligible for enrollment.)
* AHI >50 on any PSG or portable sleep study.
* Mean nocturnal heart rate > 80 bpm on baseline PSG will exclude from randomization.
* Patients receiving, narcotics or benzodiazepines unless on stable doses.
* Current alcohol or narcotic abuse as documented in the patient medical record.
* Inability or unwillingness to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the electrophysiology service of the VAPHS for CRT implant are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Shalaby, MD, Principal Investigator — VA Pittsburgh Healthcare System
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Shalaby A, Atwood CW, Selzer F, Suffoletto M, Gorcsan Iii J, Strollo P. Cardiac resynchronization therapy and obstructive sleep-related breathing disorder in patients with congestive heart failure. Pacing Clin Electrophysiol. 2011 May;34(5):593-603. doi: 10.1111/j.1540-8159.2010.03015.x. PMID 21609340